CLINICAL TRIAL: NCT04241042
Title: Clinical Validation of the Bordeaux Maze Test
Acronym: BORMATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Collaborators: Aelis Farma (Industry)
Responsible Party: Sponsor
Other Study IDs: BORMATE/2
Record Dates: First submitted 2019-11-13; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-10

CONDITIONS: Down Syndrome; Healthy
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endocannabinoid content
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Down syndrome volunteers: Males and females from 16 to 35 years
- Healthy volunteers: Males and females from 18 to 35 years

SUMMARY:
Currently, the instruments used in translational studies related to cognition have proved to be inaccurate. For this reason, the objective of this study is to evaluate whether the Bordeaux Maze Test has adequate psychometric properties and is valid for its use to compare trials tested in preclinical (animal) studies and clinical population with Down syndrome. Specifically, it is intended to study the domains of memory (relational memory) and executive functions (work memory), both relevant in the cognitive functioning of the population with Down syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome population:

  * Males and females aged 16 to 35 years.
  * Clinical diagnosis of DS (full trisomy 21 or translocated) confirmed by chromosomal analysis (karyotyping).
  * Parent or legal guardian/representative and caregiver willing to give written informed consent.
  * Study participants must have sufficient vision and hearing to participate in study evaluations. Mild hearing loss will be allowed.
  * Availability of parent/caregiver to accompany the subject to clinical visits.
  * Subjects must be able to understand basic instructions.
  * Parent or legal guardian/representative and caregiver willing to give written informed consent
* Normotypical population:

  * Males and females aged 18 to 35 years.
  * Clinical history and physical examination demonstrating no organic or psychiatric disorders.
  * Understanding and accepting the study procedures and signing the informed consent.

Exclusion Criteria:

* Study participants with a current DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) diagnosis of any primary or secondary psychiatric diagnoses (such as autism spectrum disorder, attention deficit hyperactivity disorder, depression and conduct disorder). Participation are allowed as long as they are considered stable and their medication with a regime that does not change in the 6 weeks prior to enrolment and does not interfere with the progression of the study.
* Subjects with evidence of dementia or meeting clinical diagnoses for dementia.
* Subjects thyroid dysfunction or diabetes that is not adequately controlled or stabilized on treatment for at least 8 weeks prior to randomization.
* Personal history of infantile spasms, of epilepsy, of severe head trauma or Central Nervous System (CNS) infections (e.g. meningitis), with the exception of a single isolated febrile seizure.
* Subjects with past history of seizures from primary causes (such as West syndrome and Lennox-Gastaut syndrome) or secondary causes.
* Clinical history of moderate or severe Obstructive Sleep Apnea (OSA) as defined by Apnea-Hypopnea Index (AHI) (>15 events per hour not well controlled by positive airway pressure therapy with stable settings) for at least 3 months prior to screening visit.
* Alcohol and/or substance use disorder in the past year.
* Concomitant disease or condition or any clinically significant finding at screening that could interfere with the conduct of the study, or that would, in the opinion of the investigator, could lead to an unacceptable risk to the subject in this study.
* Participation in other clinical trials in the last 3 months prior to the study.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Down syndrome volunteers are recruited from Down syndrome foundations and control volunteers from educational centres nearby the research institute.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Validation of the Bordeaux Maze Test | Changes from months 0 to months 1 and 3
  To validate a novel neuropsychological test, the Bordeaux Maze Test for the evaluation of working memory in subjects with Down syndrome (DS)

SECONDARY OUTCOMES:
Test retest reliability | months 0, 1 and 3
  To validate the Bordeaux Maze Test, for the evaluation of cognitive flexibility in subjects with Down syndrome (DS)
Criteria validity | months 0, 1 and 3
  To evaluate the influence of age and gender on the Bordeaux Maze Test in the Down syndrome population;
Analyses of the stability: Learning and practice effects observe on the Bordeaux Maze Test | months 0, 1 and 3
  To evaluate the relevance of learning/practice effects
Analyses of the stability: Learning and practice effects observe on the NIH Toolbox | months 0, 1 and 3
  To evaluate the relevance of learning/practice effects
Analyses of the stability: Floor/ ceiling effects on the Bordeaux Maze Test | months 0, 1 and 3
  To evaluate the relevance of floor/ceiling effects
Analyses of the stability: Floor/ ceiling effects on the NIH Toolbox | months 0, 1 and 3
  To evaluate the relevance of floor/ceiling effects

CONTACTS AND LOCATIONS:
Locations (1):
- IMIM (Institut Hospital del Mar d'Investigacions Mèdiques), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No